CLINICAL TRIAL: NCT05871086
Title: The Effect of Coenzyme Q10 Supplementation on the Clinical Outcome of Juvenile Idiopathic Arthritis Patients
Brief Title: Coenzyme Q10 in Juvenile Idiopathic Arthritis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nourhan Elsherif (Other)
Responsible Party: Sponsor-Investigator, Nourhan Elsherif, Clinical Pharmacy Master's Candidate, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACUCFPASURHDIRB2020110301#169
Record Dates: First submitted 2023-05-14; First posted 2023-05-23 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant
Masking Description: Placebo will be given to patients in the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coenzyme Q10 Group (Experimental): Patients will receive their JIA standard treatment plus 100 mg Coenzyme Q10 capsules daily for 3 months.
  Interventions: Dietary Supplement: Coenzyme Q10; Drug: Standard Regimen
- Control Group (Placebo Comparator): Patients will receive their standard JIA treatment plus placebo
  Interventions: Other: Placebo; Drug: Standard Regimen

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Coenzyme Q10 soft gelatin capsules daily for 3 months
  Arms: Coenzyme Q10 Group
Other: Placebo — Placebo Capsules
  Arms: Control Group
Drug: Standard Regimen — Patients may be receiving any of these commonly used JIA treatments including:
  * Ibuprofen - 30 to 40 mg/kg/day in 3 to 4 divided doses
  * Diclofenac - 2 to 3 mg/kg/day in divided doses 2 to 3 times daily
  * Methotrexate - Initial: 10 to 15 mg/m2 once weekly; adjust gradually up to 20 to 30 mg/m2 once weekly
  * Leflunomide - Weight based, 10-20 mg once daily
  * Sulfasalazine - 30 to 50 mg/kg/day in 2 divided doses
  * Etanercept - 0.8 mg/kg/dose once weekly
  * Adalimumab - Weight based, 10-40 mg every other week

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatological disorder in childhood of unknown cause and a major cause of functional disability. Standard JIA treatment including nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroids, methotrexate, and biological agents have considerable adverse effects in addition to their high cost. Despite the success of these treatment approaches, patients may still have active disease with other sequelae from chronic inflammation and considerable morbidity that may negatively impact patients' quality of life. Therefore, evaluating the potential benefit of alternative add-on anti-inflammatories and antioxidants might be a promising area for further research. Coenzyme Q10 (CoQ10) is a natural mitochondrial electron carrier and a powerful lipophilic antioxidant located in almost all cell membranes and plasma lipoproteins. Several preclinical studies in animal models as well as clinical trials in adult patients with rheumatoid arthritis (RA) have demonstrated the beneficial effects of CoQ10. Results show that CoQ10 can reduce the oxidative and inflammatory status as well as clinical features that characterize this systemic autoimmune disease.

Also, CoQ10 has been used safely in children before and was well tolerated. Thus, the investigators would like to evaluate the effect of CoQ10 oral supplementation in pediatric JIA patients.

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatological disorder in childhood of unknown etiology and a major cause of functional disability. It has a prevalence rate of about 1/1000 worldwide. The American College of Rheumatology (ACR) defines JIA as inflammation in one or more joints of unknown etiology with onset prior to age 16 years and a minimum of 6 weeks duration, following the exclusion of other known causes of synovitis. The International League of Associations for Rheumatology criteria classifies JIA into several different subgroups depending on the number of joints affected, presence of extra-articular manifestations such as uveitis or glomerulonephritis, systemic symptoms, serology and genetic factors. Peripheral arthritis is the common predominant clinical presentation among the various types. The three main types of JIA are polyarticular, oligoarticular, and systemic JIA. Therefore, diagnosis of JIA depends on physical findings, medical history, and the exclusion of other diagnoses.

The main hallmark of JIA is joint inflammation with bone resorption and tissue destruction.

This chronic inflammation limits the daily activities and productivity of patients. Interleukin-1 (IL-1), IL-6, IL-17, and tumor necrosis factor-α (TNF-α) are inflammatory cytokines that play an important role in the pathogenesis, prognosis, disease activity, and systemic features of JIA. Additionally, abnormal activation of T-cells, B-cells, natural killer (NK) cells, dendritic cells (DC), macrophages and neutrophils contribute to the pathogenesis of JIA.

All medications used to treat JIA including nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroids, methotrexate, and biological agents have considerable adverse effects in addition to the high cost of the biologics. Also, despite the success of these treatment approaches, patients may still have active disease with other sequelae from chronic inflammation and considerable morbidity that may negatively impact patients' quality of life. Therefore, evaluating the potential benefit of alternative add-on anti-inflammatories and antioxidants might be a promising area for further research.

Coenzyme Q10 (CoQ10) is a mitochondrial electron carrier and a powerful lipophilic antioxidant located in almost all cell membranes and plasma lipoproteins. It can be found naturally and acquired from the diet or synthesized in-vivo by all cells of the body. Various in-vitro and animal studies have demonstrated the antioxidant and anti-inflammatory effect of CoQ10.7 This has raised interest in its therapeutic potential against pathologies related to mitochondrial dysfunction and enhanced oxidative stress such as systemic autoimmune diseases.

Several preclinical studies in animal models as well as clinical trials in patients with rheumatoid arthritis (RA) have demonstrated the beneficial effects of CoQ10. Results show that CoQ10 can reduce the oxidative and inflammatory status as well as clinical features that characterize this systemic autoimmune disease.

In an attempt to understand the mechanisms by which CoQ10 exerts its anti-inflammatory and immunomodulatory effect, Jhun et al conducted two studies on induced-arthritis mice models. Their results showed that the mice that received CoQ10 showed significant decrease in RA severity. Immunohistochemical analysis of synovial tissue showed that CoQ10 administration lead to significantly lower levels of proinflammatory cytokines such as IL-21, IL-1, IL-6, IL-17, TNF-α and vascular endothelial growth factor (VEGF). Also, oxidative stress markers including nitrotyrosine and inducible nitric oxide synthase (iNOS) expression were significantly reduced in mice treated with CoQ10. CoQ10 also exhibited immunomodulatory effects on B and T-cells, such as down-regulating IL-17 expression and Th17 cells population induced by inflammatory response.

Furthermore Bauerova et al. exhibited that the addition of CoQ10 to methotrexate (MTX), the most commonly prescribed anti-rheumatic agent, suppressed the progression of RA in rats more than MTX alone. The effect on oxidative stress and immunomodulation was shown through a decrease in the plasma levels of MDA and IL-1, respectively.10 CoQ10 also proved that it has a protective role against hepatotoxicity caused by methotrexate. This effect was shown in a study by Tawfik et al. where liver function enzymes improved after the combination of CoQ10 with MTX in rats.

To further elucidate the effect of CoQ10 supplementation, two randomized clinical trials tested its use in adult rheumatoid arthritis patients. Abdollahzad et al. focused on the effect of CoQ10 on oxidative stress and inflammatory markers. They registered a significant decrease in serum levels of MDA & TNF-α, and trending decrease in IL-6. Moreover, no adverse drug events were observed confirming the safety and tolerability of CoQ10. With more focus on disease activity, Nachvak et al reported significant decrease in Disease Activity Scores (DAS-28), swollen joint count, tender joint count, and the visual analogue scale (VAS) scores accompanied by a reduction in erythrocyte sedimentation rate (ESR) and matrix metalloproteinase (MMP-3) levels.

Altogether, evidence supports the beneficial effect of CoQ10 supplementation not only on inflammatory markers and oxidative stress but also on clinical features and presentation of arthritis patients. Also, CoQ10 has been used in doses up to 20 mg/kg/day in children safely and was well tolerated. Up to date, there is no published study to evaluate the use of CoQ10 in JIA. Thus, the investigators would like to evaluate the effect of CoQ10 oral supplementation as adjuvant therapy on the clinical outcomes in pediatric JIA patients.

A prospective, randomized, controlled, single blind clinical trial will be conducted on 60 Juvenile Idiopathic Arthritis (JIA) patients at the Pediatric Allergy, Immunology, Rheumatology Clinic, Children's Hospital, Ain Shams University.

At baseline, caregivers of patients who are eligible will be educated about the study protocol and will be required to sign a written informed consent before enrollment in the study.

Sixty patients will be recruited in the study and will be randomized to one of the following groups:

A) Intervention (Coezyme Q10) Group (30 patients): will receive their JIA standard treatment plus 100 mg Coenzyme Q10 capsules daily for 3 months.

B) Control Group (30 patients): will receive their standard JIA treatment plus placebo

Blood samples will be withdrawn from patients at baseline and at the end of the 3 months trial period. After 3 months of CoQ10 supplementation, all the outcomes will be reassessed and reported to determine the effect on CoQ10 supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (<16 years old)
* Diagnosed with active JIA according to the American College of Rheumatology (ACR) 2019 guideline.
* Patients with peripheral oligo or polyarthritis.
* With more than 6-month disease duration
* Participants who have inadequate response to at least one first line standard therapy.
* Patients who have been receiving a stable treatment regimen for the past 3 months

Exclusion Criteria:

* Patients with active systemic JIA
* Patients presenting with complications (such as amyloidosis, uveitis, or glomerulonephritis)
* Patients with other chronic autoimmune disease.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Evaluation | 3 months
  Clinical efficacy will be assessed by calculating the Clinical Juvenile Arthritis Disease Activity Score (cJADAS-10) at baseline and at the end of the 3-month trial period.
  The cJADAS is computed by assessing the following variables:
  1. Physician's global rating of overall disease activity
  2. Parent/child ratings of well-being
  3. Counts of active joints assessed in 10 joints

SECONDARY OUTCOMES:
Serum Malondialdehyde | 3 months
  an oxidative stress markers, Malondialdehyde (MDA) will be assessed form patients sera at baseline and after 3 months. It will be measured using ELISA Kits
Serum Tumor necrosis factor-alpha | 3 months
  serum samples will be withdrawn from each patient at baseline and after 3 months . Tumor necrosis factor-alpha will be measured using an ELISA Kit.
Safety of Coenzyme Q10 | 3 months
  CoQ10 safety will be monitored by asking the parents through interviews and phone calls every 2 weeks about the occurrence of any of the following side effects: abdominal discomfort, loose stools, headache, nausea, and vomiting. assessment will be done every 2 weeks
The Childhood Health Assessment Questionnaire (CHAQ) | 3 months
  The Childhood Health Assessment Questionnaire (CHAQ) assesses functional ability in 8 domains of physical function (30 items) for children (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities). Each item is scored on a four-point scale ranging from 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), 3 (unable to do). The mean score of the eight domains finally makes up the disability index and ranges from 0 (no disability) to 3 (disabled).
  Quality of life scores will be performed for patients at baseline and at the end of the 3-months trial period.
serum glutathione | 3 months
  an oxidative stress markers, glutathione will be assessed form patients sera at baseline and after 3 months. It will be measured using ELISA Kits

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Allergy, Immunology, Rheumatology Clinic, Children's Hospital, Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prakken B, Albani S, Martini A. Juvenile idiopathic arthritis. Lancet. 2011 Jun 18;377(9783):2138-49. doi: 10.1016/S0140-6736(11)60244-4. PMID 21684384
- [Background] Giancane G, Consolaro A, Lanni S, Davi S, Schiappapietra B, Ravelli A. Juvenile Idiopathic Arthritis: Diagnosis and Treatment. Rheumatol Ther. 2016 Dec;3(2):187-207. doi: 10.1007/s40744-016-0040-4. Epub 2016 Aug 12. PMID 27747582
- [Background] Zaripova LN, Midgley A, Christmas SE, Beresford MW, Baildam EM, Oldershaw RA. Juvenile idiopathic arthritis: from aetiopathogenesis to therapeutic approaches. Pediatr Rheumatol Online J. 2021 Aug 23;19(1):135. doi: 10.1186/s12969-021-00629-8. PMID 34425842
- [Background] Ringold S, Angeles-Han ST, Beukelman T, Lovell D, Cuello CA, Becker ML, Colbert RA, Feldman BM, Ferguson PJ, Gewanter H, Guzman J, Horonjeff J, Nigrovic PA, Ombrello MJ, Passo MH, Stoll ML, Rabinovich CE, Schneider R, Halyabar O, Hays K, Shah AA, Sullivan N, Szymanski AM, Turgunbaev M, Turner A, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Treatment of Juvenile Idiopathic Arthritis: Therapeutic Approaches for Non-Systemic Polyarthritis, Sacroiliitis, and Enthesitis. Arthritis Care Res (Hoboken). 2019 Jun;71(6):717-734. doi: 10.1002/acr.23870. Epub 2019 Apr 25. PMID 31021516
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Bentinger M, Tekle M, Dallner G. Coenzyme Q--biosynthesis and functions. Biochem Biophys Res Commun. 2010 May 21;396(1):74-9. doi: 10.1016/j.bbrc.2010.02.147. PMID 20494114
- [Background] Lopez-Pedrera C, Villalba JM, Patino-Trives AM, Luque-Tevar M, Barbarroja N, Aguirre MA, Escudero-Contreras A, Perez-Sanchez C. Therapeutic Potential and Immunomodulatory Role of Coenzyme Q10 and Its Analogues in Systemic Autoimmune Diseases. Antioxidants (Basel). 2021 Apr 13;10(4):600. doi: 10.3390/antiox10040600. PMID 33924642
- [Background] Jhun J, Moon J, Ryu J, Shin Y, Lee S, Cho KH, Kang T, Cho ML, Park SH. Liposome/gold hybrid nanoparticle encoded with CoQ10 (LGNP-CoQ10) suppressed rheumatoid arthritis via STAT3/Th17 targeting. PLoS One. 2020 Nov 6;15(11):e0241080. doi: 10.1371/journal.pone.0241080. eCollection 2020. PMID 33156836
- [Background] Jhun J, Lee S, Kim SY, Na HS, Kim EK, Kim JK, Jeong JH, Park SH, Cho ML. Combination therapy with metformin and coenzyme Q10 in murine experimental autoimmune arthritis. Immunopharmacol Immunotoxicol. 2016;38(2):103-12. doi: 10.3109/08923973.2015.1122619. Epub 2015 Dec 17. PMID 26681425
- [Background] Bauerova K, Paulovicova E, Mihalova D, Drafi F, Strosova M, Mascia C, Biasi F, Rovensky J, Kucharska J, Gvozdjakova A, Ponist S. Combined methotrexate and coenzyme Q(1)(0) therapy in adjuvant-induced arthritis evaluated using parameters of inflammation and oxidative stress. Acta Biochim Pol. 2010;57(3):347-54. Epub 2010 Sep 9. PMID 20827446
- [Background] Tawfik MK. Combination of coenzyme Q10 with methotrexate suppresses Freund's complete adjuvant-induced synovial inflammation with reduced hepatotoxicity in rats: Effect on oxidative stress and inflammation. Int Immunopharmacol. 2015 Jan;24(1):80-7. doi: 10.1016/j.intimp.2014.11.018. Epub 2014 Dec 3. PMID 25488045
- [Background] Nachvak SM, Alipour B, Mahdavi AM, Aghdashi MA, Abdollahzad H, Pasdar Y, Samadi M, Mostafai R. Effects of coenzyme Q10 supplementation on matrix metalloproteinases and DAS-28 in patients with rheumatoid arthritis: a randomized, double-blind, placebo-controlled clinical trial. Clin Rheumatol. 2019 Dec;38(12):3367-3374. doi: 10.1007/s10067-019-04723-x. Epub 2019 Aug 7. PMID 31392559
- [Background] Abdollahzad H, Aghdashi MA, Asghari Jafarabadi M, Alipour B. Effects of Coenzyme Q10 Supplementation on Inflammatory Cytokines (TNF-alpha, IL-6) and Oxidative Stress in Rheumatoid Arthritis Patients: A Randomized Controlled Trial. Arch Med Res. 2015 Oct;46(7):527-33. doi: 10.1016/j.arcmed.2015.08.006. Epub 2015 Sep 3. PMID 26342738
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Miyamae T, Seki M, Naga T, Uchino S, Asazuma H, Yoshida T, Iizuka Y, Kikuchi M, Imagawa T, Natsumeda Y, Yokota S, Yamamoto Y. Increased oxidative stress and coenzyme Q10 deficiency in juvenile fibromyalgia: amelioration of hypercholesterolemia and fatigue by ubiquinol-10 supplementation. Redox Rep. 2013;18(1):12-9. doi: 10.1179/1351000212Y.0000000036. PMID 23394493
- [Background] Consolaro A, Negro G, Chiara Gallo M, Bracciolini G, Ferrari C, Schiappapietra B, Pistorio A, Bovis F, Ruperto N, Martini A, Ravelli A. Defining criteria for disease activity states in nonsystemic juvenile idiopathic arthritis based on a three-variable juvenile arthritis disease activity score. Arthritis Care Res (Hoboken). 2014 Nov;66(11):1703-9. doi: 10.1002/acr.22393. PMID 24980508
- [Background] Consolaro A, Ruperto N, Bazso A, Pistorio A, Magni-Manzoni S, Filocamo G, Malattia C, Viola S, Martini A, Ravelli A; Paediatric Rheumatology International Trials Organisation. Development and validation of a composite disease activity score for juvenile idiopathic arthritis. Arthritis Rheum. 2009 May 15;61(5):658-66. doi: 10.1002/art.24516. PMID 19405003
- [Background] Singh G, Athreya BH, Fries JF, Goldsmith DP. Measurement of health status in children with juvenile rheumatoid arthritis. Arthritis Rheum. 1994 Dec;37(12):1761-9. doi: 10.1002/art.1780371209. PMID 7986222
- [Background] el Miedany YM, Youssef SS, el Gaafary M. Cross cultural adaptation and validation of the Arabic version of the Childhood Health Assessment Questionnaire for measuring functional status in children with juvenile idiopathic arthritis. Clin Exp Rheumatol. 2003 May-Jun;21(3):387-93. PMID 12846063